CLINICAL TRIAL: NCT04270929
Title: Pressure Enabled Drug Delivery By Pancreatic Retrograde Venous Infusion For Advanced Pancreatic Carcinoma
Acronym: PANC-001
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: Roger Williams Medical Center (Other)
Collaborators: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Principal Investigator, Ritesh Rathore, MD, Director, Division of Hematology/Oncology, Roger Williams Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 342-30
Record Dates: First submitted 2020-01-16; First posted 2020-02-17 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Unresectable Pancreatic Cancer; Metastatic Pancreatic Cancer; Oxaliplatin; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — IFL protocol; folfirinox

STUDY DESIGN:
Intervention Model Description: This is an open label, single institution, single-arm, dose-escalation phase 1 study, designed to assess the feasibility, safety, and efficacy of oxaliplatin PEDD-PRVI with systemic FOLFIRI followed by FOLFIRINOX therapy for the treatment of patients with unresectable or metastatic pancreatic adenocarcinoma
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Oxaliplatin PEDD-PRVI (Experimental): Two infusions of oxaliplatin (dose escalation: 20-40 mg) over the course of 4 weeks by Pancreatic Retrograde Venous Infusion (PRVI) utilizing Pressure Enabled Drug Delivery (PEDD) technology.
  Interventions: Drug: FOLFIRI; Drug: FOLFIRINOX; Device: TriSalus Infusion System

INTERVENTIONS:
Drug: FOLFIRI — During Cycles 1 and 2, standard of care systemic FOLFIRI will be delivered on Days 2-4 following oxaliplatin PEDD-PRVI.
Drug: FOLFIRINOX — During Cycles 3-6, standard of care systemic FOLFIRINOX will be administered on Days 1-3.
Device: TriSalus Infusion System — The TriSalus Infusion System administers therapeutics using PEDD technology.

SUMMARY:
This is an open label, single institution, dose-escalation phase 1 study designed to assess the feasibility, safety, and efficacy of oxaliplatin administered via Pancreatic Retrograde Venous Infusion (PRVI) using Pressure Enabled Drug Delivery (PEDD) technology. Oxaliplatin PEDD-PRVI is administered with systemic FOLFIRI followed by FOLFIRINOX therapy for the treatment of patients with unresectable or metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
The treatment period consists of 6 cycles. Cycles 1 and 2 involve the regional administration of oxaliplatin via PEDD-PRVI with systemic FOLFIRI. During cycles 1 and 2, patients are evaluated on days 1, 2, 4, and 8. Cycles 3 through 6 include the systemic administration of standard of care FOLFIRINOX. During cycles 3 through 6, patients are evaluated on days 1 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed diagnosis of adenocarcinoma of the pancreas. Patient must have either histologic confirmation of the primary tumor or metastasis.
* Patients must have locally advanced, unresectable or metastatic pancreatic adenocarcinoma.
* Patient must be between 18 - 80 years of age.
* Patient able to understand and sign informed consent.
* Patient may be chemotherapy naïve or may have failed one line of conventional therapy
* Prior FOLFIRINOX therapy:

  * Patients who have previously received FOLFIRINOX chemotherapy for locally advanced unresectable pancreatic cancer are eligible for enrollment upon this study if they meet the following criteria-

    1. FOLFIRINOX chemotherapy was completed more than six months ago,
    2. Patients who are currently candidates for re-challenge with FOLFIRINOX chemotherapy for their recurrent cancer, and
    3. Patients have no persistent non-hematologic toxicity greater than grade 1 (due to prior FOLFIRINOX therapy)
  * Patients with metastatic cancer who are currently receiving FOLFIRINOX chemotherapy are eligible for enrollment upon this study if they meet the following criteria-

    1. Patients have received no more than six cycles of FOLFIRINOX chemotherapy,
    2. Patients have at least stable disease on imaging, and
    3. Patients have no persistent non-hematologic toxicity greater than grade 1 (due to ongoing FOLFIRINOX therapy)
* Patient with a life expectancy of greater than six months.
* Patient with performance status of 0 to 1 (ECOG).
* All patients must have adequate organ function as defined by:

  * ANC greater than or equal to 1500/mm3, platelets ≥ 100,000/mm3, Hgb ≥ to 8 g/dL; patient may be transfused to achieve Hgb ≥ 8 g/dL to satisfy enrollment criteria, or as otherwise indicated by symptoms for Hgb > 8 g/dL.
  * Creatinine ≤ 1.5mg/dl or creatinine clearance ≤ 60cc/min.
  * Direct bilirubin <1.5X ULN, alkaline phosphatase <5X ULN, and ALT/AST <5X ULN (ULN = upper limit of normal).
  * No evidence of congestive heart failure, symptoms of coronary artery disease, serious cardiac arrhythmias, including uncontrolled atrial fibrillation/atrial flutter, evidence of prior myocardial infarction by history or EKG.
  * No serious, symptomatic obstructive or emphysematous lung disease, or asthma requiring intravenous medications within the past 12 months; no serious lung disease associated with dyspnea at normal activity levels (grade III) or at rest (grade IV), due to any cause (including cancer metastases and pleural effusions).
* Acceptable vascular anatomy as determined by CT, MR, or conventional venography.

Exclusion Criteria:

* Female patients of childbearing age will be tested for pregnancy. Pregnant and breastfeeding patients will be excluded from the study. Males who are actively seeking to have children will be made aware of the unknown risks of this study protocol on human sperm and the need to practice birth control.
* Patients with serious or unstable renal, hepatic, pulmonary, cardiovascular, endocrine, rheumatologic, or allergic disease based on history, physical exam and laboratory tests will be excluded.
* Patients with uncontrolled diabetes mellitus or a history of pancreatitis.
* Patients with cholelithiasis and a history of choledocholithiasis.
* Patients with concurrent malignancies, except for cutaneous carcinomas.
* Patients with unsuitable vascular anatomy.
* Portal vein occlusion/thrombosis, history of portal hypertension, cirrhosis, hepatitis, or with radiographic evidence of cirrhosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Completion Rate of oxaliplatin PEDD-PRVI | 3 months
  To determine the completion rate of oxaliplatin delivery by PEDD-PRVI as measured by the percentage of successful placements of the TriSalus Infusion System and delivery of the assigned dose of oxaliplatin regionally into the pancreas via RVI per each patient, at each dose-level, and across all enrolled patients in the study. Successful delivery of oxaliplatin by PEDD-PRVI will be confirmed using real-time fluoroscopic guidance. The success rate of completion of PEDD-RVI per patient and acroos all-patients will be calculated
Safety of oxaliplatin PEDD-PRVI: maximum tolerable dose (MTD) | 3 months
  To determine the safety of oxaliplatin PEDD-PRVI by identifying the maximum tolerable dose (MTD).

SECONDARY OUTCOMES:
To determine local progression free survival | 3 months
  Assess the time frame of pancreatic tumor stability prior to progression by radiographic imaging
To determine systemic progression free survival. | 3 months
  Assess the time frame of metastatic tumor stability prior to progression by radiographic imaging
To determine overall survival | 3 months
  As a measure of activity, overall survival will be assessed. The events for the assessment of overall survival are death events.
Radiographic response rates by PET | 3 months
  Changes in tumor metabolic activity
Radiographic response rate by perfusion MRI | 3 months
  Changes in tumor size
Serologic response rates (CA 19-9) | 3 months
  Serial measurement of serum CA 19-9 levels

CONTACTS AND LOCATIONS:
Overall Officials: Rathore, Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No